CLINICAL TRIAL: NCT01597310
Title: An Open-Label Study to Assess the Effect of Dexpramipexole (BIIB050) on the Pharmacokinetics of Warfarin in Healthy Volunteers
Brief Title: Dexpramipexole and Warfarin Drug Drug Interaction (DDI) Study
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Knopp Biosciences (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Basic Science
Other Study IDs: 223HV105
Record Dates: First submitted 2012-05-10; First posted 2012-05-14 (Estimated); Last update posted 2014-11-25 (Estimated); Status verified 2014-11

CONDITIONS: Healthy Volunteers
MeSH Terms: interventions — Warfarin; Dexpramipexole

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Warfarin (Experimental): 25 mg Warfarin, Treatment Period 1 & Treatment Period 2
  Interventions: Drug: Warfarin
- Dexpramipexole (Experimental): 150 mg BID Treatment Period 2
  Interventions: Drug: Dexpramipexole

INTERVENTIONS:
Drug: Warfarin — single doses at specified time periods
  Arms: Warfarin
Drug: Dexpramipexole — multiple doses
  Arms: Dexpramipexole

SUMMARY:
This study will assess the effect of dexpramipexole on the pharmacokinetics (PK) of the CYP2C9 probe substrate warfarin in healthy volunteers.

DETAILED DESCRIPTION:
This is a single center open label study to assess the effect of Dexpramipexole on the PK of Warfarin in Healthy Volunteers. The goals of this study are as follows: to assess the effect of dexpramipexole on the pharmacodynamics (PD) of warfarin, to assess the safety and tolerability of dexpramipexole when administered alone, and with warfarin, and to assess the PK of dexpramipexole when administered alone; to explore the influence of genetic variation on the PK and international normalized ratio (INR) of warfarin when administered alone, and with dexpramipexole; and to explore the influence of genetic variation on the PK of dexpramipexole when administered alone.

ELIGIBILITY:
Inclusion Criteria:

* Subjects who, in the opinion of the investigator, are healthy as determined by medical history, physical examination, and 12 Lead ECG.
* Adult males/females aged 18 to 55 years inclusive.
* Male and female subjects of childbearing age must practice effective contraception during the study and up to 90 days after their last dose of study drug.

Exclusion Criteria:

* History of malignant disease, including solid tumors and hematologic malignancies.
* Clinically significant current active infection or serious infection.
* History of gastrointestinal bleeding, peptic ulcer disease, hemorrhoids or epistaxis.
* Personal or family history of any bleeding disorder, and/or coagulation profile results outside of normal limits.
* Known allergy or hypersensitivity to warfarin.

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 15 (Actual)
Dates: Start 2012-05; Primary Completion 2012-07 (Actual); Study Completion 2012-07 (Actual)

PRIMARY OUTCOMES:
Determination of the effect of dexpramipexole on the pharmacokinetics (PK) parameters of the CYP2C9 probe substrate warfarin including: AUC: area under the plasma-concentration time curve over a specified time period and Cmax: Maximum observed plasma c | pre-dose and at 0.5, 1, 2, 3, 4, 6, 8, 12, 24, 48, 72, 96 and 144 hours after warfarin administration in each dosing period
PK parameters of dexpramipexole including but not limited to AUC: area under the plasma-concentration time curve over a specified time period and Cmax: Maximum observed plasma concentration | pre-dose and at 0.25, 0.5, 0.75, 1, 1.5, 2, 2.5, 3, 4, 6, 8 and 12 hours after administration of the morning dexpramipexole dose on Day 1 and Day 12 of Period 2

CONTACTS AND LOCATIONS:
Locations (1):
- Research Site, Overland Park, Kansas, United States